CLINICAL TRIAL: NCT03392116
Title: A Phase 1 Randomized, Double Blind, Placebo Controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NGM120 in Healthy Adult Subjects
Brief Title: Single and Multiple Ascending Dose Study of NGM120 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0401
Record Dates: First submitted 2017-12-08; First posted 2018-01-05 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: NGM120 (Experimental): Single Dose
  Interventions: Biological: NGM120
- Part A: Placebo (Placebo Comparator): Single Dose
  Interventions: Other: Placebo
- Part B: NGM120 (Experimental): Multiple Dose
  Interventions: Biological: NGM120
- Part B: Placebo (Placebo Comparator): Multiple Dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM120 — Subcutaneous Injection
  Arms: Part A: NGM120; Part B: NGM120
Other: Placebo — Subcutaneous Injection
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose is to evaluate the safety, tolerability, and PK of NGM120 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Normal ECG findings

Exclusion Criteria:

* Significant history or clinical manifestation of any allergic, dermatological, hepatic, renal, hematological, pulmonary, metabolic, cardiovascular, gastrointestinal, neurological, or psychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Part A Arm-Single Dose: Treatment Emergent Adverse events | 28 days
  Percentage of total subjects with Treatment Emergent Adverse event
Part B Arm-Multiple Dose: Treatment Emergent Adverse events | 84 days
  Percentage of total subjects with Treatment Emergent Adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Limited, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No